CLINICAL TRIAL: NCT01650480
Title: HELPing Older People With Very Severe Chronic Obstructive Pulmonary Disease (COPD) Towards the End of Their Lives: Developing, Piloting and Refining a Practical Intervention (HELP-COPD)
Brief Title: HELPing Older People With Very Severe Chronic Obstructive Pulmonary Disease Towards the End of Their Lives: Developing, Piloting and Refining a Practical Intervention (HELP-COPD)
Acronym: HELP-COPD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: The Dunhill Medical Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012/R/RES/02; 12243 (Registry Identifier: UKCRN ID)
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2014-02-12 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; holistic; pilot; intervention
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: HELP-COPD action plan
- Control group (No Intervention)

INTERVENTIONS:
Other: HELP-COPD action plan — The trial specialist nurse trained in palliative aspects of respiratory care will arrange a meeting to suit the patients' clinical condition and convenience. During the meeting the HELP-COPD action plan will be worked through by the patient and study nurse, and any areas of concern will be identified. Based on the findings of the assessment, a range of actions points may be generated. All referrals will be made through the usual channels. Issues that have arisen from the assessment will be clearly recorded on the HELP-COPD action plan and by ensuring that all agencies and the patient have copies of the plan it is hoped that the planned action points will be reviewed and implementation facilitated. The action plan will be reviewed by the study nurse who will contact the patient at 1, 3 and 6 months to check progress with action points.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to develop, refine and pilot a novel complex (HELP-COPD) assessment, undertaken during or immediately after a hospital admission, which addresses the holistic care needs of people with severe chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Registered with Lothian General Practice
* Admitted with an exacerbation of COPD as their primary diagnosis at Royal Infirmary of Edinburgh

Exclusion Criteria:

* People with lung cancer
* People unable to give informed consent and complete questionnaire booklets in English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
FACIT | 3 and 6 months
  The Functional Assessment of Chronic Illness Therapy (FACIT) measurement system has a core of 27 validated questions in four domains: Physical, Social/Family, Emotional, and Functional well-being. Scores range from 0 (worst quality of life) to 108, and are responsive to change with a minimum clinically important difference for improvement of 5.5. A sub-scale of 10 questions for use in lung cancer is considered to be appropriate in other respiratory conditions.

SECONDARY OUTCOMES:
The St George Respiratory Questionnaire (SGRQ) | 3 and 6 months
MRC Dyspnoea score | 3 and 6 months
Dyspnoea 12 | 3 and 6 months
COPD Assessment Test (CAT) | 3 and 6 months
The Hospital Anxiety and Depression Scale (HADS) | 3 and 6 months
FACIT Spiritual Well-Being sub-scale (FACIT-Sp) | 3 and 6 months
Palliative care Outcome Scale (POS) | 3 and 6 months
EQ-5D | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Pinnock, Dr, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, City of Edinburgh, United Kingdom

REFERENCES:
- [Derived] Kendall M, Buckingham S, Ferguson S, MacNee W, Sheikh A, White P, Worth A, Boyd K, Murray SA, Pinnock H. Exploring the concept of need in people with very severe chronic obstructive pulmonary disease: a qualitative study. BMJ Support Palliat Care. 2018 Dec;8(4):468-474. doi: 10.1136/bmjspcare-2015-000904. Epub 2015 Aug 26. PMID 26310525
- See also: HELP-COPD — http://www.cphs.mvm.ed.ac.uk/projects/help-copd/